CLINICAL TRIAL: NCT05913388
Title: Randomized Double-Blind Placebo Controlled Phase II Study of a Galectin-3 Inhibitor (GB1211) and Pembrolizumab Versus Pembrolizumab and Placebo in Patients With Metastatic Melanoma and Head and Neck Squamous Cell Carcinoma
Brief Title: GB1211 and Pembrolizumab Versus Pembrolizumab and Placebo in Patients With Metastatic Melanoma and Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center (Unknown); Providence Cancer Center, Earle A. Chiles Research Institute (Other); Galecto Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023000353
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma; Head and Neck Squamous Cell Carcinoma
Keywords: metastatic melanoma; head and neck squamous cell carcinoma; pembrolizumab; galecto; GB1211
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GB1211 + Pembrolizumab (Experimental): GB1211 will be administered orally twice a day at 400mg in combination with standard pembrolizumab treatment.
  Interventions: Drug: GB1211; Drug: Pembrolizumab
- Pembrolizumab Monotherapy (Placebo Comparator): Placebo will have the same appearance as GB1211 and administered orally twice a day in combination with standard pembrolizumab treatment.
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: GB1211 — Administered orally twice daily at 100mg.
  Arms: GB1211 + Pembrolizumab
Drug: Pembrolizumab — Administered at a fixed dose of 200 mg every 3 weeks intravenously.
  Other Names: Keytruda
Drug: Placebo — Administered orally twice daily at 100mg.
  Arms: Pembrolizumab Monotherapy

SUMMARY:
The purpose of this study is to determine the objective response of GB1211 and pembrolizumab versus pembrolizumab and placebo in patients with advance metastatic melanoma or head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Eligible patients will be registered, stratified by diagnosis (melanoma versus oral, head and neck (OHN) cancer), and the number of prior systemic therapies, and randomized to receive either GB1211 + pembrolizumab or pembrolizumab + placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic melanoma including unknown primary or mucosal melanomas. Histological confirmation of melanoma will be required by previous biopsy or cytology. Patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) with disease progression during or after platinum-containing chemotherapy are eligible. PD-L1 testing is not needed for OHN cancers.
* Patients who have received anti-PD1 or anti-PD-L1 in the past are eligible if it has been at least 6 months since the last anti-PD-1 or PD-L1 dose, they meet all other eligibility criteria and progression of malignancy has been documented on imaging. Progression for this patient subset is defined as the appearance of one or more new metastatic sites, or a 5% or greater increase in the sum of diameter of target lesions or an unequivocal increase in non-target site. Treatment naïve melanoma patients are eligible.
* Patients must be ≥ 18 years of age.
* ECOG performance status of 0-2.
* Women of childbearing potential must have a serum or urine pregnancy test performed within 72 hours prior to the start of protocol treatment. The results of this test must be negative in order for the patient to be eligible. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy.
* No active bleeding.
* Anticipated lifespan greater than 12 weeks.
* Patients must sign a study-specific consent document.

Exclusion Criteria:

* Patients who have previously received a galectin antagonist.
* Patients with active autoimmune disease except for autoimmune thyroiditis or vitiligo.
* Patients with history of autoimmune colitis.
* Patients with untreated brain metastases. Patients with treated brain metastases who demonstrate control of brain metastases with follow-up imaging 4 or more weeks after initial therapy are eligible.
* Patients requiring other systemic oncologic therapy, including experimental therapies.
* Patients who have received anti-cancer treatment within 3 weeks or 5 half-lives before first study drug dose.
* Patients with Child-Pugh C hepatic impairment.
* Patients with active infection requiring antibiotics.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Need for steroids at greater than physiologic replacement doses. Inhaled corticosteroids are acceptable.
* Laboratory exclusions (to be performed within 28 days of enrollment):

  * WBC < 3.0 x 109/L
  * Hgb < 9.0 g/dL
  * AST or ALT > 1.5 times ULN
  * Total bilirubin > 1.9 g/dL, unless due to Gilbert's Syndrome. If Gilbert's Syndrome is present by clinical history, then direct bilirubin must by < 3.0 g/dl.
  * Active or known history of HIV
  * Active or known history of Hepatitis B
  * Active or known history of Hepatitis C
  * Platelet counts < 100 x 10E9 / L (100,000/ μL) without transfusion
  * INR > 1.5x ULN
* Inability to give informed consent and comply with the protocol. Patients must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.
* Any medical condition that in the opinion of the Principal Investigator would compromise the safety or conduct of the study procedures.
* Unresolved immune-mediated pneumonitis, diarrhea, elevation of hepatocellular enzymes or other toxicities requiring greater than physiological replacement doses of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Overall response rate based on disease imaging | From the date of randomization until the date of first documented progression, assessed up to 63 weeks.
  Determine the response of Gal-3 inhibitor and pembrolizumab versus pembrolizumab monotherapy (plus placebo) in patients with metastatic melanoma or head and neck squamous cell carcinoma (HNSCC).

SECONDARY OUTCOMES:
Evaluation of GAL-3 Expression | Screening and Day 68
  Compare Gal-3 expression in paired biopsies after GB1211 + pembrolizumab or pembrolizumab monotherapy
Evaluation of Predictive Biomarker | Day 85
  Characterize myeloid-derived suppressor cells (MDSC) expression over time as a predictive biomarker of response after GB1211 + pembrolizumab or pembrolizumab monotherapy
Frequency of Immune-mediated Adverse Events | From the time of informed consent to week 63
  Compare the frequency of immune-mediated adverse events after GB1211 + pembrolizumab versus pembrolizumab + placebo
Evaluation of Antiviral Immunity | Day 85
  Assess the biological activity of GB1211 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring CD4+T cells with a memory phenotype (CD3+CD4+Ki67+CD25+FoxP3-CCR7-CD45RA-CD27+CD28+/-).
Evaluation of Antiviral Immunity | Day 85
  Assess the biological activity of GB1211 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring CD8+ T cells with effector phenotype (CD3+CD8+CD28-CD95+).
Evaluation of Antiviral Immunity | Day 85
  Assess the biological activity of GB1211 + pembrolizumab and in comparison to pembrolizumab monotherapy by measuring tumor-specific T cells using autologous and/or HLA-matched tumor when available.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan D. Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT05913388/ICF_000.pdf